CLINICAL TRIAL: NCT01687231
Title: A Randomized Pilot Study Comparing Infection Rates in Myeloablative Allogeneic Stem Cell Transplant Patients Receiving a Non-Neutropenic Diet or a Neutropenic Diet
Brief Title: Infection Rates of Myeloablative Allo SCT Recipients Receiving Neutropenic Diets Versus Non-Neutropenic Diets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00012374; Pro00012374 (Other: DUHS IRB)
Record Dates: First submitted 2012-09-11; First posted 2012-09-18 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Hematologic Malignancies
Keywords: Neutropenic Diet, Non-Neutropenic Diet, Allogeneic SCT
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neutropenic Diet (No Intervention): This arm is the control and subjects will receive the standard of care neutropenic diet.
- Non-neutropenic Diet (Experimental): This arm is interventional and subjects will receive a non-neutropenic diet without restriction.
  Interventions: Other: Non-neutropenic Diet

INTERVENTIONS:
Other: Non-neutropenic Diet — Non-neutropenic diet is without restriction.
  Arms: Non-neutropenic Diet

SUMMARY:
In the transplant community, there is debate regarding the most appropriate food services for stem cell transplant patients. Recommendations regarding the use of low bacterial diets have been based on theoretical concepts of reducing the risk of contracting infections from pathogens found in food sources rather than clinical trials. The evidence for the use of a neutropenic diet is weak. To date, there have been little to no randomized controlled studies addressing the question whether a neutropenic diet in addition to prophylactic antibiotics is necessary as infection prevention in myeloablative stem cell transplant patients. For this reason, our research is aimed at providing data to substantiate the use of neutropenic diets in preventing infections in recipients of myeloablative stem cell transplants.

DETAILED DESCRIPTION:
In the proposed pilot study, a randomized design will be used to address the primary and secondary aims. Subjects will be randomized to either the experimental group receiving a non-neutropenic diet without restriction, or to the control group receiving the standard neutropenic diet. While randomization will occur prior to, or on the day of their inpatient admission and the subjects will begin study procedures upon admission to the Adult Stem Cell Transplant Inpatient Unit at Duke University Medical Center.

The diet will continue until 1) the subject is no longer neutropenic, and/or 2) discharged from the inpatient unit to continue their care in the Adult Stem Cell Transplant Outpatient Clinic. By limiting the study to the time of care on the inpatient unit, we will minimize the opportunity for deviation from the assigned diet. Absence of neutropenia will be defined as an absolute neutrophil count of greater than 500/uL (manual differential) and a total white blood cell count of 1000/uL for three consecutive days.

All subjects enrolled will follow the standard prophylactic antibiotic regimen. Other supportive care will also be consistent in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo a myeloablative allogeneic stem cell transplant for any cancer or non-cancer illness from any related or unrelated donor source including bone marrow, peripheral blood progenitor cell, or umbilical cord blood
2. Age 20-70 years of age
3. Karnofsky Performance Scale KPS> 80
4. Ability to read and write English

Exclusion Criteria:

1. Autologous stem cell transplant recipients
2. Non-myeloablative or reduced intensity stem cell transplant recipients
3. Pregnant women
4. Patients with a documented active infection prior to starting their preparative regimen. This includes grade 3 or higher viral, bacterial, or fungal infection.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Bacteremia | Duration of hospitalization or neutropenia, an expected average of 5 weeks.
  Participants will be followed for the duration of hospital stay or until neutropenic, an expected average of 5 weeks. The time frame will be measured from the date of randomization until the date of discharge from the inpatient unit of the hospital or until they are assessed to be neutropenic, whichever came first, assessed up to 8 weeks.

SECONDARY OUTCOMES:
Assess nutritional status using PG-SGA | Duration of hospitalization or neutropenia, an expected average of 5 weeks.
  The participants will be followed for the duration of hospital stay or until neutropenic, an expected average of 5 weeks. The time frame will measured from the date of randomization until the date of discharge from the inpatient unit of the hospital or until they are assessed to be neutropenic, whichever came first, assessed up to 8 weeks. The nutritional status will be assessed by the Scored Patient-Generated Subjective Global Assessment (PG-SGA) platform.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Chao, MD, MBA, Study Chair — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States